CLINICAL TRIAL: NCT01485757
Title: Effect of Chronic Oral L-arginine Supplementation on Peripheral Endothelial Function and Exercise Tolerance in a Population of Young Heart Transplant Patients.
Brief Title: Prospective L-arginine Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Technical difficulty with Endo-PAT machine
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Josh Friedland-Little, MD, Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00035716
Record Dates: First submitted 2011-11-29; First posted 2011-12-05 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Heart Transplant
Keywords: patients
MeSH Terms: interventions — Arginine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- L-arginine (Experimental)
  Interventions: Drug: L-arginine

INTERVENTIONS:
Drug: L-arginine — All study subjects will be treated with a 12 week (11-13 week) course of oral L-arginine at a dose of 6 g per day, divided into morning and evening doses of 3 g (3 1000 mg capsules or caplets).

SUMMARY:
HYPOTHESIS The investigators primary hypothesis is that peripheral endothelial function and exercise tolerance will be abnormal in the population of young heart transplant patients at baseline, and that each will show a trend towards improvement following a 12 week course of oral L-arginine, with regression towards the baseline following the 12 week washout period.

ELIGIBILITY:
Inclusion Criteria:

* University of Michigan Pediatric Heart Transplant Clinic patient.
* Greater than or equal to 8 years of age.
* Heart transplant between 1 and 8 years prior to enrollment in the study

Exclusion Criteria:

* Relative hypotension for age
* Refusal to participate
* Inability to cooperate with Endo-PAT testing
* Pregnant or nursing women.
* Insulin dependent diabetes

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in peripheral endothelial function from baseline following 12 week treatment course of L-arginine. | baseline and 12 weeks
  Endothelial function will be assessed at baseline as well as after a 12 week treatment course of L-arginine. A final measurement will be made following a 12 week washout period.

SECONDARY OUTCOMES:
Change from baseline in serum levels of oxidative stress markers | baseline and 12 weeks
  Serum markers of oxidative stress will be measured at baseline and after a 12 week treatment course of L-arginine. A final measurement will be made after a 12 week washout period.
Change in exercise tolerance from baseline following a 12 week treatment course of L-arginine | baseline and 12 weeks
  Exercise tolerance will be assessed with a 6 minute walk at baseline and following a 12 week treatment course of L-arginine. A final measurement will be made after a 12 week washout period.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Pediatric Heart Transplant Clinic, Ann Arbor, Michigan, United States